CLINICAL TRIAL: NCT00360698
Title: Comparison of Two Therapeutic Strategies for Treating Type 2 Diabetic Patients Poorly Controlled With Basal Insulin Associated With Oral Antidiabetic Drugs : 6-month Proof of Concept Study.
Brief Title: Insulin Glulisine in Type 2 Diabetic Patients
Acronym: Basal Plus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMR1964A_4002; EUDRACT # : 2005-002614-38
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Results first posted 2009-12-02 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; glimepiride; insulin glulisine; Metformin

ARMS (2):
- insulin glulisine+insulin glargine+metformin+glimepiride (Other): Bolus arm
  Interventions: Drug: Insulin Glargine; Drug: Glimepiride; Drug: Insulin Glulisine; Drug: Metformin
- insulin glargine+metformin+glimepiride (Other): Control arm
  Interventions: Drug: Insulin Glargine; Drug: Glimepiride; Drug: Metformin

INTERVENTIONS:
Drug: Insulin Glargine — One daily injection at bedtime
Drug: Glimepiride — At same dosage as during the run-in period
Drug: Insulin Glulisine — One bolus given before the main meal
  Arms: insulin glulisine+insulin glargine+metformin+glimepiride
Drug: Metformin — At same dosage as during the run-in period

SUMMARY:
To evaluate the efficacy of a single injection of glulisine before the main meal added to insulin glargine plus oral antidiabetic drugs (OADs) compared to insulin glargine plus OADs in Type 2 diabetic patients poorly controlled with basal insulin plus OADs.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus, Type 2
* 25 < BMI < 45 kg/m²
* 7,5% < HbA1c < 9%
* Treated with a basal insulin (NPH, Insulin Zinc, Insulin glargine or Insulin detemir), and at least 1g metformin daily, for more than 3 months

Exclusion Criteria:

* Type 1 diabetes mellitus
* Treatment with OADs only
* Treatment with thiazolidinediones, with exenatide or with pramlintide
* Treatment with an insulin other than basal insulin (Premix, rapid insulin, fast-acting insulin analogue)
* Active proliferative diabetic retinopathy,
* Pregnancy (women of childbearing potential must have a negative pregnancy test at study entry and effective contraception)
* Breast-feeding
* History of hypersensitivity to the study drugs or to drugs with a similar chemical structure.
* Treatment with systemic corticosteroids in the 3 months prior to study entry
* Treatment with any investigational product in the 2 months prior to study entry
* Previous treatment with insulin glulisine
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol
* Clinically relevant cardiovascular, hepatic, neurological, endocrine, or other major disease making implementation of the protocol or interpretation of the study results difficult
* Impaired hepatic function
* Impaired renal function
* History of drug or alcohol abuse

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2006-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: PILORGET Valérie, MD, Study Director — Sanofi
Locations (3):
- Sanofi-aventis, Bridgewater, New Jersey, United States
- Sanofi-Aventis, Moscow, Russia
- Sanofi-aventis, Guildford, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During Run-In period patients were not assigned to a treatment group. They were all treated with Insulin Glargine + Metformin + Glimepiride.
Groups:
- Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride: Insulin Glulisine (One daily injection at main meal) + Insulin Glargine (One daily injection at bedtime) + Metformin (At same dosage as during the run-in period) + Glimepiride (At same dosage as during the run-in period)
- Insulin Glargine+Metformin+Glimepiride: Insulin Glargine (One daily injection at bedtime) + Metformin (At same dosage as during the run-in period) + Glimepiride (At same dosage as during the run-in period)
Period: Run-In
Arm/Group | Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride | Insulin Glargine+Metformin+Glimepiride
Started | 0 | 135
Completed | 0 | 125 (19 patients completed the run-in but were not eligible for randomization in the treatment period)
Not Completed | 0 | 10
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Non compliance with treatment procedure | 0 | 1
Not completed — Sponsor request | 0 | 2
Not completed — Patient did not meet inclusion criteria | 0 | 1
Not completed — Patient personal reasons | 0 | 2
Not completed — Need of insulin with meals | 0 | 1
Period: Treatment Period
Arm/Group | Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride | Insulin Glargine+Metformin+Glimepiride
Started | 49 | 57
Completed | 48 | 56
Not Completed | 1 | 1
Not completed — Non compliance with treatment procedure | 1 | 0
Not completed — Early termination by error | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride | Insulin Glargine+Metformin+Glimepiride | Total
Number analyzed (Participants) | 49 | 57 | 106
Age Continuous [Mean (Standard Deviation); unit: years] | 60.6 (6.73) | 59.3 (8.84) | 59.9 (7.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 35 | 64
  Male | 20 | 22 | 42
Region of Enrollment [Number; unit: participants]
  United States | 23 | 27 | 50
  United Kingdom | 11 | 14 | 25
  Russian Federation | 15 | 16 | 31
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] — Total patients analyzed n=105 due to one missing data in the "insulin glulisine+insulin glargine+metformin+glimepiride" group
  kg/m² | 33.2 (5.30) | 33.3 (4.39) | 33.3 (4.80)
Daily Mean Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] — Patients having a baseline value and a value on treatment:
  insulin glulisine+insulin glargine+metformin+glimepiride group n=47 patients, insulin glargine+metformin+glimepiride group n=55 patients
  mg/dL | 170.2 (27.86) | 167.4 (39.41) | 169 (34.33)
Duration of diabetes [Mean (Standard Deviation); unit: years] | 12.1 (7.29) | 11.0 (7.02) | 11.5 (7.13)
Glycosylated Haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percent] | 7.8 (0.60) | 8.0 (0.67) | 7.9 (0.64)
Weight [Mean (Standard Deviation); unit: kg] — Total patients analyzed n=105 due to one missing data in the "insulin glulisine+insulin glargine+metformin+glimepiride" group
  kg | 91.5 (16.60) | 92.9 (17.15) | 92.3 (16.83)

OUTCOME MEASURES:

1. Primary Outcome: Patients With Glycosylated Haemoglobin (HbA1c) Value < 7%
Description: Glycosylated Haemoglobin (HbA1c) is a biological parameter that reflects the blood glucose concentration over a long period of time. It is the standard parameter for glycemic control follow -up in diabetic patients. this parameter is expressed in percentage (%) and the target in diabetes management is to reach a HbA1c <7%
Time Frame: at the end of treatment (week 24)
Population: Modified Intent to treat (ITT) population, LOCF (Last Observation Carried Forward)
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride | Insulin Glargine+Metformin+Glimepiride
Number analyzed (Participants) | 49 | 57
percentage of participants | 22.4 | 8.8
Statistical Analysis 1: Comparison: Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride vs Insulin Glargine+Metformin+Glimepiride; The null-hypothesis stated no differences between the 2 treatment groups regarding the percentage of patients with Glycosylated Haemoglobin (HbA1c) level <7%. A sample size of 98 randomized (49/arm) patients would allow to demonstrate with 80% power that 40 % of patients in the Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride group would achieve a HbA1c level < 7 % compared to 15 % of patients in the Insulin Glargine+Metformin+Glimepiride group(5% alpha risk, 2-sided test); Test type: Superiority or Other; p = 0.0499, Chi-squared; Risk Difference (RD) = 13.68, 95% CI [0.01 to 28.37] — Difference in percentage between groups: Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride group - Insulin Glargine+Metformin+Glimepiride group

2. Secondary Outcome: Glycosylated Haemoglobin (HbA1c) Value
Time Frame: at the end of treatment (week 24)
Population: Modified ITT population, LOCF
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride | Insulin Glargine+Metformin+Glimepiride
Number analyzed (Participants) | 49 | 57
percent | 7.5 (0.64) | 7.8 (0.85)

3. Secondary Outcome: Change in Glycosylated Haemoglobin (HbA1c) Value
Time Frame: from baseline to the end of treatment (week 24)
Population: Modified ITT population, LOCF
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride | Insulin Glargine+Metformin+Glimepiride
Number analyzed (Participants) | 49 | 57
percent | -0.37 (0.085) | -0.11 (0.078)
Statistical Analysis 1: Comparison: Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride vs Insulin Glargine+Metformin+Glimepiride; The null-hypothesis stated no difference between the 2 treatment groups regarding the adjusted mean change from baseline in Glycosylated Haemoglobin (HbA1c) at the end of treatment; Test type: Superiority or Other; p = 0.029, ANCOVA — Threshold for statistical significance (alpha) = 0.05 ; 2 sided-test; The analysis is an ANCOVA analysis on the change with group as fixed effect and baseline HbA1c as covariate; Mean Difference (Net) = -0.26, 95% CI [-0.49 to -0.03], Standard Error of Mean 0.116 — Difference between groups: Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride group - Insulin Glargine+Metformin+Glimepiride group

4. Secondary Outcome: Daily Mean Plasma Glucose
Time Frame: at the end of treatment (week 24)
Population: Modified ITT population, LOCF
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride | Insulin Glargine+Metformin+Glimepiride
Number analyzed (Participants) | 47 | 55
mg/dL | 154.7 (28.62) | 165.8 (37.48)

5. Secondary Outcome: Change in Daily Mean Plasma Glucose
Time Frame: from baseline to the end of treatment (week 24)
Population: Modified ITT population, LOCF
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride | Insulin Glargine+Metformin+Glimepiride
Number analyzed (Participants) | 47 | 55
mg/dL | -15.01 (3.661) | -2.07 (3.384)
Statistical Analysis 1: Comparison: Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride vs Insulin Glargine+Metformin+Glimepiride; The null-hypothesis stated no differences between the 2 treatment groups regarding the adjusted mean change from baseline in daily mean plasma glucose at the end of treatment; Test type: Superiority or Other; p = 0.0109, ANCOVA — Threshold for statistical significance (alpha) = 0.05 ; 2 sided-test; The analysis is an ANCOVA analysis on the change with group as fixed effect and baseline daily mean plasma glucose as covariate; Mean Difference (Net) = -12.94, 95% CI [-22.83 to -3.04], Standard Error of Mean 4.987 — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: Change in Weight
Time Frame: from baseline to the end of treatment (week 24)
Population: Modified ITT population, LOCF
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride | Insulin Glargine+Metformin+Glimepiride
Number analyzed (Participants) | 48 | 56
kg | 0.46 (0.316) | 0.22 (0.293)
Statistical Analysis 1: Comparison: Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride vs Insulin Glargine+Metformin+Glimepiride; The null-hypothesis stated no differences between the 2 treatment groups regarding the adjusted mean change from baseline in weight at the end of treatment; Test type: Superiority or Other; p = 0.5762, ANCOVA — Threshold for statistical significance (alpha) = 0.05 ; 2 sided-test; The analysis is an ANCOVA analysis on the change with group as fixed effect and baseline weight as covariate; Mean Difference (Net) = 0.24, 95% CI [-0.61 to 1.1], Standard Error of Mean 0.431 — [estimate comment as in outcome 3, analysis 1]

7. Secondary Outcome: Daily Dose of Insulin Glargine
Description: Mean of 3 daily doses reported during the week prior to the final visit
Time Frame: at the end of treatment (week 24)
Population: Modified ITT population, LOCF
Measure: Mean (Standard Deviation); unit: units of insulin glargine per day
Arm/Group | Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride | Insulin Glargine+Metformin+Glimepiride
Number analyzed (Participants) | 49 | 57
units of insulin glargine per day | 54.7 (34.84) | 62.2 (34.85)

8. Secondary Outcome: Daily Dose of Insulin Glulisine
Description: Mean of 3 daily doses reported during the week prior to the final visit
Time Frame: at the end of treatment (week 24)
Population: Modified ITT population, LOCF
Measure: Mean (Standard Deviation); unit: units of insulin glulisine per day
Arm/Group | Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride | Insulin Glargine+Metformin+Glimepiride
Number analyzed (Participants) | 49 | 0
units of insulin glulisine per day | 12.8 (6.59) |

9. Secondary Outcome: Rate of Symptomatic Hypoglycemia With Plasma Glucose < 70mg/dL
Time Frame: during treatment period (12 weeks)
Population: Safety population
Measure: Mean (Standard Deviation); unit: Number of hypoglycemia per patient-year
Arm/Group | Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride | Insulin Glargine+Metformin+Glimepiride
Number analyzed (Participants) | 49 | 57
Number of hypoglycemia per patient-year | 8.19 (14.603) | 7.68 (13.996)
Statistical Analysis 1: Comparison: Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride vs Insulin Glargine+Metformin+Glimepiride; The null-hypothesis stated no difference between the 2 treatment groups regarding the rate of symptomatic hypoglycemia with plasma glucose <70 mg/dL during the treatment period; Test type: Superiority or Other; p = 0.958, Wilcoxon (Mann-Whitney) — Threshold for statistical significance (alpha) = 0.05 ; 2 sided-test

10. Secondary Outcome: Rate of Nocturnal Symptomatic Hypoglycemia With Plasma Glucose < 70mg/dL
Time Frame: during treatment period (12 weeks)
Population: Safety population
Measure: Mean (Standard Deviation); unit: Number of hypoglycemia per patient-year
Arm/Group | Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride | Insulin Glargine+Metformin+Glimepiride
Number analyzed (Participants) | 49 | 57
Number of hypoglycemia per patient-year | 1.62 (3.418) | 3.95 (9.339)
Statistical Analysis 1: Comparison: Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride vs Insulin Glargine+Metformin+Glimepiride; The null-hypothesis stated no difference between the 2 treatment groups regarding the rate of nocturnal symptomatic hypoglycemia with plasma glucose <70 mg/dL during the treatment period; Test type: Superiority or Other; p = 0.302, Wilcoxon (Mann-Whitney) — Threshold for statistical significance (alpha) = 0.05 ; 2 sided-test

11. Secondary Outcome: Rate of Severe Symptomatic Hypoglycemia
Time Frame: during treatment period (12 weeks)
Population: Safety population
Measure: Mean (Standard Deviation); unit: Number of hypoglycemia per patient-year
Arm/Group | Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride | Insulin Glargine+Metformin+Glimepiride
Number analyzed (Participants) | 49 | 57
Number of hypoglycemia per patient-year | 0.00 (0.000) | 0.20 (1.096)
Statistical Analysis 1: Comparison: Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride vs Insulin Glargine+Metformin+Glimepiride; The null-hypothesis stated no difference between the 2 treatment groups regarding the rate of severe symptomatic hypoglycemia during the treatment period; Test type: Superiority or Other; p = 0.192, Wilcoxon (Mann-Whitney) — Threshold for statistical significance (alpha) = 0.05 ; 2 sided-test

ADVERSE EVENTS:
Arm/Group | Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride | Insulin Glargine+Metformin+Glimepiride
Serious Adverse Events (participants affected / at risk) | 1/49 | 2/57
Other Adverse Events (participants affected / at risk) | 0/49 | 0/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Insulin Glulisine+Insulin Glargine+Metformin+Glimepiride (N=49) | Insulin Glargine+Metformin+Glimepiride (N=57)
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendon Disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.